CLINICAL TRIAL: NCT00039364
Title: Open Label Phase II Study On STI571 (Glivec) Administered As A Daily Oral Treatment In Gliomas
Brief Title: Imatinib Mesylate in Treating Patients With Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16011-26013; EORTC-16011; EORTC-26013
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult pilocytic astrocytoma; adult subependymoma; adult giant cell glioblastoma; adult gliosarcoma; adult diffuse astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Glioma, Subependymal; Gliosarcoma | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may interfere with the growth of tumor cells and slow the growth of the tumor.

PURPOSE: Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic activity of imatinib mesylate (in terms of objective response and progression-free survival at 6 months) in patients with gliomas.
* Determine the safety of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to glioma (glioblastoma multiforme vs anaplastic oligodendroglioma or mixed oligoastrocytoma vs anaplastic astrocytoma or recurrent low-grade astrocytoma).

Patients receive oral imatinib mesylate once or twice daily. Treatment repeats every 4 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 6 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 77 patients (29 patients with glioblastoma multiforme, 24 patients with anaplastic oligodendroglioma or mixed oligoastrocytoma, and 24 patients with anaplastic astrocytoma or recurrent low-grade astrocytoma) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed glioblastoma multiforme

  * Recurrent disease by CT scan or MRI
  * No prior chemotherapy OR
  * No more than 1 prior chemotherapy regimen in adjuvant setting or for recurrent disease OR
* Histologically or cytologically confirmed anaplastic oligodendroglioma, mixed oligoastrocytoma, anaplastic astrocytoma, or recurrent low-grade astrocytoma

  * Failed prior radiotherapy
  * No more than 1 prior chemotherapy regimen

    * Failed adjuvant chemotherapy OR
    * Failed first-line chemotherapy
* At least 1 bidimensionally measurable target lesion

  * At least 2 cm on contrast-enhanced CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine less than 1.7 mg/dL

Cardiovascular:

* Cardiac function normal
* No ischemic heart disease within the past 6 months
* Normal 12-lead ECG

Other:

* No other prior or concurrent malignancy except cone-biopsied carcinoma of the cervix or adequately treated basal cell or squamous cell skin cancer
* No unstable systemic disease
* No active uncontrolled infection
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent anticancer biologic agents
* No concurrent cytokines (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea)
* No concurrent chemotherapy

Endocrine therapy:

* Must be on stable or decreasing dose of corticosteroids for at least 2 weeks

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior brain irradiation
* No prior high-dose radiotherapy (more than 65 Gy), stereotactic radiosurgery, or internal radiotherapy unless the recurrence is histologically confirmed
* No concurrent radiotherapy

Surgery:

* Prior surgery for primary brain tumor within the past 3 months allowed provided one of the following conditions are present:

  * Postoperative imaging within 72 hours after surgery shows a clearly limited target lesion of at least 2 cm
  * Postoperative follow-up shows a progressive and measurable target lesion
  * A second measurable target lesion is present outside the surgical area

Other:

* No concurrent warfarin or other anticoagulants
* No other concurrent anticancer agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-03; Primary Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Raymond, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Martin J. van Den Bent, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (10):
- Kaiser Franz Josef Hospital, Vienna, Austria
- U.Z. Gasthuisberg, Leuven, Belgium
- France (4):
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Institut Gustave Roussy, Villejuif
- Azienda Ospedaliera di Padova, Padua, Italy
- Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam, Netherlands
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Beatson Oncology Centre, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Raymond E, Brandes AA, Dittrich C, Fumoleau P, Coudert B, Clement PM, Frenay M, Rampling R, Stupp R, Kros JM, Heinrich MC, Gorlia T, Lacombe D, van den Bent MJ; European Organisation for Research and Treatment of Cancer Brain Tumor Group Study. Phase II study of imatinib in patients with recurrent gliomas of various histologies: a European Organisation for Research and Treatment of Cancer Brain Tumor Group Study. J Clin Oncol. 2008 Oct 1;26(28):4659-65. doi: 10.1200/JCO.2008.16.9235. PMID 18824712
- [Result] Raymond E, Brandes A, Van Oosterom A, et al.: Multicentre phase II study of imatinib mesylate in patients with recurrent glioblastoma: an EORTC: NDDG/BTG Intergroup study. [Abstract] J Clin Oncol 22 (Suppl 14): A-1501, 2004.